CLINICAL TRIAL: NCT05350163
Title: Phase I Dose Escalation of T-cell Receptor α/β Depleted Donor Lymphocyte Infusions Following CD34+- Selected Allogeneic Stem Cell Transplantation From Related & Unrelated Donors in Patients With Lymphoid, Myeloid or Plasma Cell Malignancies
Brief Title: T-cell Receptor α/β Depleted Donor Lymphocyte Infusion
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study met criteria for stopping due to lack of efficacy per protocol specifications.
Sponsor: Guenther Koehne (Other)
Responsible Party: Sponsor-Investigator, Guenther Koehne, Deputy Director and Chief of Blood and Marrow Transplant, Hematologic Oncology and Benign Hematology, Baptist Health South Florida
Organization: Baptist Health South Florida (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KOE-004
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lymphoid Leukemia, Acute; Myeloid Malignancy; Plasma Cell Tumor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Plasmacytoma

STUDY DESIGN:
Intervention Model Description: The model is both parallel and sequential, in that Matched and Mismatched strata run in parallel and independently. Within each stratum, Cohorts I-III are filled sequentially. In addition, Cohort I of each stratum has three groups (A-C) that are filled sequentially.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- HLA Matched Cohort I (Experimental): 5 x 10^5/kg at 6-7 weeks post-transplant (Group A), 4-5 weeks post-transplant (Group B), or 2-3 weeks post-transplant (Group C)
  Interventions: Biological: T-cell Receptor α/β Depleted Donor Lymphocyte Infusions
- HLA Matched Cohort II (Experimental): 5 x 10^5/kg starting time point X (whichever was safest as determined by Matched Cohort I), 1 x 10^6/kg 3-4 weeks after first dose, and 1 x 10^6/kg 3-4 weeks after second dose
  Interventions: Biological: T-cell Receptor α/β Depleted Donor Lymphocyte Infusions
- HLA Matched Cohort III (Experimental): 5 x 10^5/kg starting time point X (whichever was safest as determined by Matched Cohort I), 1 x 10^6/kg 3-4 weeks after first dose, and 2 x 10^6/kg 3-4 weeks after second dose
  Interventions: Biological: T-cell Receptor α/β Depleted Donor Lymphocyte Infusions
- HLA Mismatched Cohort I (Experimental): 1 x 10^5/kg at 6-7 weeks post-transplant (Group A), 4-5 weeks post-transplant (Group B), or 2-3 weeks post-transplant (Group C)
  Interventions: Biological: T-cell Receptor α/β Depleted Donor Lymphocyte Infusions
- HLA Mismatched Cohort II (Experimental): 1 x 10^5/kg starting time point Y (whichever was safest as determined by Mismatched Cohort I), 5 x 10^5/kg 3-4 weeks after first dose, and 5 x 10^5/kg 3-4 weeks after second dose
  Interventions: Biological: T-cell Receptor α/β Depleted Donor Lymphocyte Infusions
- HLA Mismatched Cohort III (Experimental): 1 x 10^5/kg starting time point Y (whichever was safest as determined by Mismatched Cohort I), 5 x 10^5/kg 3-4 weeks after first dose, and 1 x 10^6/kg 3-4 weeks after second dose
  Interventions: Biological: T-cell Receptor α/β Depleted Donor Lymphocyte Infusions

INTERVENTIONS:
Biological: T-cell Receptor α/β Depleted Donor Lymphocyte Infusions — T-cell Receptor α/β Depleted Donor Lymphocyte Infusions following CD34+-selected Allogeneic Stem Cell Transplantation from Related and Unrelated Donors for Patients

SUMMARY:
This pilot study is being conducted to treat patients who have a certain type of malignancy (lymphoid or myeloid) with immune effector cells after a T-cell depleted allogeneic hematopoietic cell transplantation (TCD HSCT).

This study is designed to see whether an investigational cellular product of immune cells obtained from a donor's cells that have been treated so that the type of cells that can lead to graft vs host disease have been removed can be safely administered. These cell products are administered following the initial stem cell transplant to assess the effect and improvement on minimal residual disease status, infectious complication, progression-free and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies that are candidates CD34+ selected, T-cell depleted allogeneic hematopoietic stem cell transplantation.
* Patients must have a Karnofsky (adult) Performance Status of at least 70%.
* Patients must have adequate organ function measured by:

  * Cardiac: asymptomatic or if symptomatic then left ventricular ejection fraction (LVEF) at rest must be 50% and must improve with exercise.
  * Hepatic: < 3x upper limit of normal (ULN) AST and < 1.5 mg/dL total serum bilirubin, unless there is congenital benign hyperbilirubinemia. Patients with higher bilirubin levels due to causes other than active liver disease is also eligible with Pl approval (e.g., patients with PNH, Gilbert's disease or other hemolytic disorders).
  * Renal: serum creatinine: ≤ 1.2 mg/dL or if serum creatinine is outside the normal range, then creatinine clearance (CrCl) > 40 mL/min (measured or calculated/estimated).
  * Pulmonary: asymptomatic or if symptomatic, diffusing capacity of the lungs for carbon monoxide (DLCO) 50% of predicted (corrected for hemoglobin).
* Each patient must be willing to participate as a research subject and must sign an informed consent form.

Exclusion Criteria:

* Patients with active acute GvHD.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Koehne, MD, PhD, Principal Investigator — Miami Cancer Institute
Locations (1):
- Miami Cancer Institute at Baptist Health, Inc, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seggewiss R, Einsele H. Immune reconstitution after allogeneic transplantation and expanding options for immunomodulation: an update. Blood. 2010 May 13;115(19):3861-8. doi: 10.1182/blood-2009-12-234096. Epub 2010 Mar 9. PMID 20215642
- [Background] Lang P, Handgretinger R. Haploidentical SCT in children: an update and future perspectives. Bone Marrow Transplant. 2008 Oct;42 Suppl 2:S54-9. doi: 10.1038/bmt.2008.285. PMID 18978746
- [Background] Reisner Y, Hagin D, Martelli MF. Haploidentical hematopoietic transplantation: current status and future perspectives. Blood. 2011 Dec 1;118(23):6006-17. doi: 10.1182/blood-2011-07-338822. Epub 2011 Sep 14. PMID 21921045
- [Background] Jagasia M, Arora M, Flowers ME, Chao NJ, McCarthy PL, Cutler CS, Urbano-Ispizua A, Pavletic SZ, Haagenson MD, Zhang MJ, Antin JH, Bolwell BJ, Bredeson C, Cahn JY, Cairo M, Gale RP, Gupta V, Lee SJ, Litzow M, Weisdorf DJ, Horowitz MM, Hahn T. Risk factors for acute GVHD and survival after hematopoietic cell transplantation. Blood. 2012 Jan 5;119(1):296-307. doi: 10.1182/blood-2011-06-364265. Epub 2011 Oct 18. PMID 22010102
- [Background] Arora M, Klein JP, Weisdorf DJ, Hassebroek A, Flowers ME, Cutler CS, Urbano-Ispizua A, Antin JH, Bolwell BJ, Boyiadzis M, Cahn JY, Cairo MS, Isola L, Jacobsohn DA, Jagasia M, Klumpp TR, Lee SJ, Petersdorf EW, Santarone S, Gale RP, Schouten HC, Spellman S, Wingard JR, Horowitz MM, Pavletic SZ. Chronic GVHD risk score: a Center for International Blood and Marrow Transplant Research analysis. Blood. 2011 Jun 16;117(24):6714-20. doi: 10.1182/blood-2010-12-323824. Epub 2011 Apr 14. PMID 21493797
- [Background] Chao NJ, Schmidt GM, Niland JC, Amylon MD, Dagis AC, Long GD, Nademanee AP, Negrin RS, O'Donnell MR, Parker PM, et al. Cyclosporine, methotrexate, and prednisone compared with cyclosporine and prednisone for prophylaxis of acute graft-versus-host disease. N Engl J Med. 1993 Oct 21;329(17):1225-30. doi: 10.1056/NEJM199310213291703. PMID 8413388
- [Background] Nash RA, Antin JH, Karanes C, Fay JW, Avalos BR, Yeager AM, Przepiorka D, Davies S, Petersen FB, Bartels P, Buell D, Fitzsimmons W, Anasetti C, Storb R, Ratanatharathorn V. Phase 3 study comparing methotrexate and tacrolimus with methotrexate and cyclosporine for prophylaxis of acute graft-versus-host disease after marrow transplantation from unrelated donors. Blood. 2000 Sep 15;96(6):2062-8. PMID 10979948
- [Background] Ratanatharathorn V, Nash RA, Przepiorka D, Devine SM, Klein JL, Weisdorf D, Fay JW, Nademanee A, Antin JH, Christiansen NP, van der Jagt R, Herzig RH, Litzow MR, Wolff SN, Longo WL, Petersen FB, Karanes C, Avalos B, Storb R, Buell DN, Maher RM, Fitzsimmons WE, Wingard JR. Phase III study comparing methotrexate and tacrolimus (prograf, FK506) with methotrexate and cyclosporine for graft-versus-host disease prophylaxis after HLA-identical sibling bone marrow transplantation. Blood. 1998 Oct 1;92(7):2303-14. PMID 9746768
- [Background] Gratwohl A, Brand R, Apperley J, Biezen Av Av, Bandini G, Devergie A, Schattenberg A, Frassoni F, Guglielmi C, Iacobelli S, Michallet M, Kolb HJ, Ruutu T, Niederwieser D; Chronic Leukemia Working Party of the European Group for Blood and Marrow Transplantation (CLWP-EBMT). Graft-versus-host disease and outcome in HLA-identical sibling transplantations for chronic myeloid leukemia. Blood. 2002 Dec 1;100(12):3877-86. doi: 10.1182/blood.V100.12.3877. PMID 12433695
- [Background] Martin PJ, Schoch G, Fisher L, Byers V, Anasetti C, Appelbaum FR, Beatty PG, Doney K, McDonald GB, Sanders JE, et al. A retrospective analysis of therapy for acute graft-versus-host disease: initial treatment. Blood. 1990 Oct 15;76(8):1464-72. PMID 2207321
- [Background] Reisner Y, Kapoor N, Kirkpatrick D, Pollack MS, Dupont B, Good RA, O'Reilly RJ. Transplantation for acute leukaemia with HLA-A and B nonidentical parental marrow cells fractionated with soybean agglutinin and sheep red blood cells. Lancet. 1981 Aug 15;2(8242):327-31. doi: 10.1016/s0140-6736(81)90647-4. PMID 6115110
- [Background] Handgretinger R, Klingebiel T, Lang P, Schumm M, Neu S, Geiselhart A, Bader P, Schlegel PG, Greil J, Stachel D, Herzog RJ, Niethammer D. Megadose transplantation of purified peripheral blood CD34(+) progenitor cells from HLA-mismatched parental donors in children. Bone Marrow Transplant. 2001 Apr;27(8):777-83. doi: 10.1038/sj.bmt.1702996. PMID 11477433
- [Background] Jakubowski AA, Small TN, Young JW, Kernan NA, Castro-Malaspina H, Hsu KC, Perales MA, Collins N, Cisek C, Chiu M, van den Brink MR, O'Reilly RJ, Papadopoulos EB. T cell depleted stem-cell transplantation for adults with hematologic malignancies: sustained engraftment of HLA-matched related donor grafts without the use of antithymocyte globulin. Blood. 2007 Dec 15;110(13):4552-9. doi: 10.1182/blood-2007-06-093880. Epub 2007 Aug 23. PMID 17717135
- [Background] Urbano-Ispizua A, Rozman C, Pimentel P, Solano C, de la Rubia J, Brunet S, Perez-Oteyza J, Ferra C, Zuazu J, Caballero D, Bargay J, Carvalhais A, Diez JL, Espigado I, Alegre A, Rovira M, Campilho F, Odriozola J, Sanz MA, Sierra J, Garcia-Conde J, Montserrat E; Spanish Group for Allogeneic Peripheral Blood Transplantation (Grupo Espanol de Trasplante Hemopoyetico) and Instituto Portugues de Oncologia-Porto. Risk factors for acute graft-versus-host disease in patients undergoing transplantation with CD34+ selected blood cells from HLA-identical siblings. Blood. 2002 Jul 15;100(2):724-7. doi: 10.1182/blood-2001-11-0057. PMID 12091376
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Devine S, Soiffer R, Pasq uini M, Carter S, Hari P, DeVore S, Stein A, Lazarus H, Linker C, Stadtrnauer E, Keever-Taylor C, O'Reil ly RJ . HLA-identical sibling matched, CD34+ selected, T cell depleted peripheral blood stem cells following rnyeloablative conditioning for first or second remission acute rnyeloid leukemia (AM L): Results of blood and marrow trans plant clinical trials network (BMT CTN) Protocol 0303. Blood, 1 14 (22), 273.
- [Background] Bethge WA, Hegenbart U, Stuart MJ, Storer BE, Maris MB, Flowers ME, Maloney DG, Chauncey T, Bruno B, Agura E, Forman SJ, Blume KG, Niederwieser D, Storb R, Sandmaier BM. Adoptive immunotherapy with donor lymphocyte infusions after allogeneic hematopoietic cell transplantation following nonmyeloablative conditioning. Blood. 2004 Feb 1;103(3):790-5. doi: 10.1182/blood-2003-07-2344. Epub 2003 Oct 2. PMID 14525766
- [Background] Peggs KS, Thomson K, Hart DP, Geary J, Morris EC, Yong K, Goldstone AH, Linch DC, Mackinnon S. Dose-escalated donor lymphocyte infusions following reduced intensity transplantation: toxicity, chimerism, and disease responses. Blood. 2004 Feb 15;103(4):1548-56. doi: 10.1182/blood-2003-05-1513. Epub 2003 Oct 23. PMID 14576063
- [Background] Frey NV, Porter DL. Graft-versus-host disease after donor leukocyte infusions: presentation and management. Best Pract Res Clin Haematol. 2008 Jun;21(2):205-22. doi: 10.1016/j.beha.2008.02.007. PMID 18503987
- [Background] Meyer RG, Britten CM, Wehler D, Bender K, Hess G, Konur A, Hartwig UF, Wehler TC, Ullmann AJ, Gentilini C, Uharek L, Huber C, Kolbe K, Herr W. Prophylactic transfer of CD8-depleted donor lymphocytes after T-cell-depleted reduced-intensity transplantation. Blood. 2007 Jan 1;109(1):374-82. doi: 10.1182/blood-2006-03-005769. Epub 2006 Aug 29. PMID 16940425
- [Background] Farhan S, Lee DA, Champlin RE, Ciurea SO. NK cell therapy: targeting disease relapse after hematopoietic stem cell transplantation. Immunotherapy. 2012 Mar;4(3):305-13. doi: 10.2217/imt.11.174. Epub 2012 Feb 13. PMID 22329587
- [Background] Handgretinger R. Negative depletion of CD3(+) and TcRalphabeta(+) T cells. Curr Opin Hematol. 2012 Nov;19(6):434-9. doi: 10.1097/MOH.0b013e3283582340. PMID 22914586
- [Background] Tyler EM, Jungbluth AA, O'Reilly RJ, Koehne G. WT1-specific T-cell responses in high-risk multiple myeloma patients undergoing allogeneic T cell-depleted hematopoietic stem cell transplantation and donor lymphocyte infusions. Blood. 2013 Jan 10;121(2):308-17. doi: 10.1182/blood-2012-06-435040. Epub 2012 Nov 16. PMID 23160468
- [Background] O'Reilly RJ, Dao T, Koehne G, Scheinberg D, Doubrovina E. Adoptive transfer of unselected or leukemia-reactive T-cells in the treatment of relapse following allogeneic hematopoietic cell transplantation. Semin Immunol. 2010 Jun;22(3):162-72. doi: 10.1016/j.smim.2010.02.003. Epub 2010 May 26. PMID 20537908
- [Background] Schumm M, Lang P, Bethge W, Faul C, Feuchtinger T, Pfeiffer M, Vogel W, Huppert V, Handgretinger R. Depletion of T-cell receptor alpha/beta and CD19 positive cells from apheresis products with the CliniMACS device. Cytotherapy. 2013 Oct;15(10):1253-8. doi: 10.1016/j.jcyt.2013.05.014. PMID 23993299
- [Background] Munchel AT, Kasamon YL, Fuchs EJ. Treatment of hematological malignancies with nonmyeloablative, HLA-haploidentical bone marrow transplantation and high dose, post-transplantation cyclophosphamide. Best Pract Res Clin Haematol. 2011 Sep;24(3):359-68. doi: 10.1016/j.beha.2011.05.001. Epub 2011 Jul 13. PMID 21925089
- [Background] Maniar A, Zhang X, Lin W, Gastman BR, Pauza CD, Strome SE, Chapoval AI. Human gammadelta T lymphocytes induce robust NK cell-mediated antitumor cytotoxicity through CD137 engagement. Blood. 2010 Sep 9;116(10):1726-33. doi: 10.1182/blood-2009-07-234211. Epub 2010 Jun 2. PMID 20519625
- [Background] Godder KT, Henslee-Downey PJ, Mehta J, Park BS, Chiang KY, Abhyankar S, Lamb LS. Long term disease-free survival in acute leukemia patients recovering with increased gammadelta T cells after partially mismatched related donor bone marrow transplantation. Bone Marrow Transplant. 2007 Jun;39(12):751-7. doi: 10.1038/sj.bmt.1705650. Epub 2007 Apr 23. PMID 17450185
- [Background] Blazar BR, Taylor PA, Bluestone JA, Vallera DA. Murine gamma/delta-expressing T cells affect alloengraftment via the recognition of nonclassical major histocompatibility complex class Ib antigens. Blood. 1996 May 15;87(10):4463-72. PMID 8639809
- [Background] Bonneville M, Scotet E. Human Vgamma9Vdelta2 T cells: promising new leads for immunotherapy of infections and tumors. Curr Opin Immunol. 2006 Oct;18(5):539-46. doi: 10.1016/j.coi.2006.07.002. Epub 2006 Jul 25. PMID 16870417
- [Background] Grimes HL, Schanie CL, Huang Y, Cramer D, Rezzoug F, Fugier-Vivier I, Ildstad ST. Graft facilitating cells are derived from hematopoietic stem cells and functionally require CD3, but are distinct from T lymphocytes. Exp Hematol. 2004 Oct;32(10):946-54. doi: 10.1016/j.exphem.2004.07.011. PMID 15504550
- [Background] Leung W. Use of NK cell activity in cure by transplant. Br J Haematol. 2011 Oct;155(1):14-29. doi: 10.1111/j.1365-2141.2011.08823.x. Epub 2011 Aug 4. PMID 21812770
- See also: Miami Cancer Institute Website — http://cancer.baptisthealth.net/miami-cancer-institute

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HLA Matched Cohort I | HLA Matched Cohort II | HLA Matched Cohort III | HLA Mismatched Cohort I | HLA Mismatched Cohort II | HLA Mismatched Cohort III
Started | 10 | 0 | 0 | 1 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated so we did not yet accrue to some cohorts, as the cohorts were filled sequentially within HLA Matched and Mismatched groupings.
Groups:
- Total: Total of all reporting groups
Arm/Group | HLA Matched Cohort I | HLA Matched Cohort II | HLA Matched Cohort III | HLA Mismatched Cohort I | HLA Mismatched Cohort II | HLA Mismatched Cohort III | Total
Number analyzed (Participants) | 10 | 0 | 0 | 1 | 0 | 0 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 0 | 0 | 1 | 0 | 0 | 6
  >=65 years | 5 | 0 | 0 | 0 | 0 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (14.3) |  |  | 57 (0) |  |  | 60.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  |  | 0 |  |  | 4
  Male | 6 |  |  | 1 |  |  | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 |  |  | 0 |  |  | 5
  Not Hispanic or Latino | 5 |  |  | 1 |  |  | 6
  Unknown or Not Reported | 0 |  |  | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0 |  |  | 0
  Asian | 0 |  |  | 1 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0 |  |  | 0
  Black or African American | 0 |  |  | 0 |  |  | 0
  White | 10 |  |  | 0 |  |  | 10
  More than one race | 0 |  |  | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 |  |  | 1 |  |  | 11

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Serious Adverse Events (TE-SAEs)
Description: TE-SAEs are defined as the composite of death, non-fatal pulmonary embolism, stroke, acute graft versus host disease (GvHD), and clinically significant laboratory test abnormalities.
Time Frame: 30 days post-infusion
Population: The study was terminated so we did not yet accrue to some cohorts, as the cohorts were filled sequentially.
Measure: Count of Participants; unit: Participants
Arm/Group | HLA Matched Cohort I | HLA Matched Cohort II | HLA Matched Cohort III | HLA Mismatched Cohort I | HLA Mismatched Cohort II | HLA Mismatched Cohort III
Number analyzed (Participants) | 10 | 0 | 0 | 1 | 0 | 0
Participants | 1 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants in Remission
Description: Remission - measured by absence of signs and symptoms
Time Frame: 2 years
Population: Because the study was terminated early, no participants completed 2 years.
Arm/Group | HLA Matched Cohort I | HLA Matched Cohort II | HLA Matched Cohort III | HLA Mismatched Cohort I | HLA Mismatched Cohort II | HLA Mismatched Cohort III
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Transplant-associated Viral Complications
Description: Transplant-associated viral complications - measured by viral infections associated with transplant
Time Frame: 2 years
Population: Because the study was terminated early, no participants completed 2 years
Arm/Group | HLA Matched Cohort I | HLA Matched Cohort II | HLA Matched Cohort III | HLA Mismatched Cohort I | HLA Mismatched Cohort II | HLA Mismatched Cohort III
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Disease Free Survival- Measured by Absence of Relapse/Recurrence or Death.
Description: Disease free survival - measured by (absence of ) relapse/recurrence or death.
  Relapse and recurrence, both will be measured by greater than 5% circulating leukemic blasts in the marrow or peripheral blood and/or the presence of blasts in any extra medullary site and/or disease determined by clinical assessment.
Time Frame: 2 years
Population: Because the study was terminated early, no participants completed 2 years.
Arm/Group | HLA Matched Cohort I | HLA Matched Cohort II | HLA Matched Cohort III | HLA Mismatched Cohort I | HLA Mismatched Cohort II | HLA Mismatched Cohort III
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival - measured by death
Time Frame: 2 years
Population: Because the study was terminated early, no participants completed 2 years.
Arm/Group | HLA Matched Cohort I | HLA Matched Cohort II | HLA Matched Cohort III | HLA Mismatched Cohort I | HLA Mismatched Cohort II | HLA Mismatched Cohort III
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The longest any participant was on study was approximately 14 months.
Description: The study was terminated so we did not yet accrue to some cohorts, as the cohorts were filled sequentially within HLA Matched and Mismatched groupings. Therefore the number of participants at risk for some groups was 0.
Arm/Group | HLA Matched Cohort I | HLA Matched Cohort II | HLA Matched Cohort III | HLA Mismatched Cohort I | HLA Mismatched Cohort II | HLA Mismatched Cohort III
All-Cause Mortality (participants affected / at risk) | 5/10 | 0/0 | 0/0 | 1/1 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 6/10 | 0/0 | 0/0 | 1/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 10/10 | 0/0 | 0/0 | 1/1 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HLA Matched Cohort I (N=10) | HLA Matched Cohort II (N=0) | HLA Matched Cohort III (N=0) | HLA Mismatched Cohort I (N=1) | HLA Mismatched Cohort II (N=0) | HLA Mismatched Cohort III (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased platelet count (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HLA Matched Cohort I (N=10) | HLA Matched Cohort II (N=0) | HLA Matched Cohort III (N=0) | HLA Mismatched Cohort I (N=1) | HLA Mismatched Cohort II (N=0) | HLA Mismatched Cohort III (N=0)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection reactivation (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other, Large B cell lymphoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased platelet count (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated ALT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated AST (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other, Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other, COVID-19 (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other, Sapovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other, Strongloidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Several of the participants had been on study for more than a year by the time the study was terminated. However, because the study was terminated early, the study did not accrue to the target, some cohorts had zero participants accrued, and no participants completed the study. Therefore, no conclusions can be drawn at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT05350163/Prot_SAP_000.pdf